CLINICAL TRIAL: NCT01233388
Title: Real-time Influenza Vaccine Surveillance: FLUNET
Brief Title: Real-time Influenza Vaccine Surveillance
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Melissa Stockwell, MD, MPH, Asst Prof of Pediatrics, Columbia University
Other Study IDs: AAAD1619
Record Dates: First submitted 2010-10-29; First posted 2010-11-03 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Vaccine Safety

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Text message surveillance: enroll for text message surveillance
  Interventions: Other: Text message surveillance

INTERVENTIONS:
Other: Text message surveillance — Text message surveillance for vaccine adverse events
  Other Names: Flunet

SUMMARY:
The aim of this proposal is to pioneer the implementation and evaluation of a novel patient centered text messaging vaccine adverse event surveillance network.

DETAILED DESCRIPTION:
The proposal will be conducted at six clinical sites of Columbia University Medical Center (CUMC), using a customized version of our already operational technology platform. Our proposed 12 month project will entail three phases: (a) 3 months of preparatory work, (b) 6 months of intervention rollout and (c) 3 months of data analysis and dissemination.

Preparatory work will include 3 areas:

Indepth interviews: We will conduct a series of interviews with patients and parents to understand their perspective on vaccine safety and Flunet. We will also interview a sample of providers to understand the most effective way for service promotion among providers. Design of registration process and messages: We will use patient/parental feedback to refine critical parts of the implementation, such as the registration process and the messages (content, frequency, format) to maximize response rates and the quality of information collected, which will be piloted in the next phase.

Technology set up and testing will occur prior to roll out in a HIPAA compliant data center. The intervention rollout will begin with a 6week refinement period. The primary goals of the refinement period are to: (1) validate/improve the methodology (e.g. registration, logic and content of the interactive menus, data collection process (2) test the application and infrastructure required for the full roll out (3) refine logistic details, such as printed materials for patients and providers. We will interview 25 patients to learn about their experience using Flunet. We will also evaluate the operations, technology and clinical findings from the intervention and incorporate any adjustments needed. After the refinement period, we will continue to monitor the systems and operations on an ongoing basis. All patients receiving a vaccine(vaccinees) will be offered the service. For children <18 years of age, a parent or guardian (parent) will be offered the service. By calling a registration number vaccinees/parents will agree to receive a series of text messages following up on the vaccinee's health.

Participating locations will include five community health centers and one hospital-based clinic, affiliated with New York Presbyterian Hospital Ambulatory Care Network (ACN) and Columbia University. These clinics include general pediatric, general medicine, Obstetric Gynecology(OBGYN)and family medicine patients. These sites are all in Health Professional Shortage Areas (HPSA).

Design and preparatory phase (months 13):

Preparatory work for implementing Flunet entails the 3 main activities: (a) Patient and provider interviews (b)Technology setup and (c) Logistic tasks.

Rollout Phase (months 39):

The roll out will entail the 3 key activities: (a) Vaccinee enrollment/registration; (b) Service delivery; (c) Refinement period and final evaluations (at 6 weeks and at the intervention end). At the beginning, we will conduct a 6 week refinement phase to validate and improve the initial design(e.g. registration methodology, best sequence and content of the interactive messages, data collection process).

The key component of the intervention is the text messaging exchange of information between our system and vaccinees. Information will comprise the following topics: (a) adverse events and (b) additional messages(primarily health tips for the influenza season). We will send a registration message and weekly messages through 6 weeks post-immunization. The first message will be sent at enrollment. Messages monitoring AEs will be sent at week 1, 2, 4, and 6, and messages containing tips and education at weeks 3 and 5. All messages detailed below are preliminary and will be modified based on feedback from vaccinees/parents obtained from the patient interviews. Messages are sent in the language selected during the telephone sign up. Additional questions will be asked only to patients reporting AEs. Messages that may trigger a reply will be designed so that vaccinees'/parents' responses are automatically parsed and replied to using a rules-based algorithm. Final messages will be based on focus group and interviews.

ELIGIBILITY:
Inclusion Criteria:

* Have an active cell phone with text messaging capability
* Presents for care at participating sites
* Fluent in English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pediatric, adult and OB patiente receiving an influenza vaccine
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2010-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Number of participants who report a health symptom within 6 weeks of vaccination | 6 weeks
  As this is a pilot study, we want to first determine if people will report health problems. Therefore, we will assess the number of participants who report a health problem within 6 weeks of vaccination.

SECONDARY OUTCOMES:
Sensitivity of the patient reporting compared to medical record | 6 weeks
  We will compare information provided by participants for moderate-to-severe health problems with the medical record to determine sensitivity of reporting.
Specificity of the patient reporting compared to medical record | 6 weeks
  We will compare information provided by participants for moderate-to-severe health problems with the medical record to determine specificity of reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Philip LaRussa, MD, Principal Investigator — Columbia University; Melissa Stockwell, MD MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States